CLINICAL TRIAL: NCT02280421
Title: A Single-centre, Open-label, Randomised, Cross-over, Drug-drug Interaction Study to Investigate the Effect of Repeated Oral Doses of Ciclosporin on the Single-dose Pharmacokinetics of nASP2151 in Healthy Mean
Brief Title: Drug-Drug Interaction Study: ASP2151 and Ciclosporin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Europe Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: M522101-EU21
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: HSV; Herpes; volunteers; drug-drug interaction; transplant
MeSH Terms: conditions — Herpes Simplex | interventions — ASP2151; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP2151 400mg (Other): ASP2151 400mg + 100mg ciclosporin
  Interventions: Drug: ASP2151 400mg + 100mg ciclosporin
- ASP2151 1200mg (Other): ASP2151 1200mg + 100mg ciclosporin
  Interventions: Drug: ASP2151 1200mg + 100mg ciclosporin

INTERVENTIONS:
Drug: ASP2151 400mg + 100mg ciclosporin
  Arms: ASP2151 400mg
Drug: ASP2151 1200mg + 100mg ciclosporin
  Arms: ASP2151 1200mg

SUMMARY:
ASP2151 is an experimental treatment for herpes. Patients undergoing organ and tissue transplantation may be prescribed ciclosporin to suppress their immune system to give the transplant an increased chance of not being rejected. A patient with a compromised immune system is more susceptible to infections such as herpes, which will require treatment.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (Quetelet index) in the range 18.0-30.9 kg/m2.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
* Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Any of the following liver function tests higher than 1.5 times the ULN at the screening visit: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), bilirubin, gamma glutamyl transpeptidase (gamma-GT).
* Platelet counts outside normal limits.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Clinically significant impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* Receipt of a live vaccine in the 3 months before the first dose of study medication, or planned immunisation with a live vaccine during the study.
* Evidence of any significant bacterial, viral, fungal or parasitic infection during the 4 weeks before dosing (minor fungal nail infections will not be regarded as significant); minor infection (eg common cold) not requiring anti-infective treatment during the 2 weeks before dosing.
* History of bleeding diathesis.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
* Presence or history of severe adverse reaction to any drug, history of multiple drug allergies (multiple defined as >3), or sensitivity to trial medication.
* Use, during the 28 days before the first dose of trial medication, of any prescription medicine, or any other medicine or herbal remedy (such as St John's wort) known to interfere with the CYP3A4 metabolic pathway (unless judged as not clinical significant by the investigator and sponsor). See Appendix 1 for common CYP3A4 interactors/substrates.
* Use, during the 7 days before the first dose of trial medication, of any over-the-counter medicine, with the exception of paracetamol (acetaminophen).
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
* Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 5 cigarettes daily.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B antigen (HBsAg); or positive test for hepatitis B core antibody (HBcAb).
* Positive test for hepatitis C, HIV1, HIV2, or active and latent tuberculosis.
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in United Kingdom from 06-October 2014 to 10-February 2015
  Each participant was randomised to 2 groups. One group was received ASP 400mg in first intervention and 1200mg in other group. There was a washout of at least 2 weeks between the interventions.
Pre-assignment Details: Participants received a single dose of 400mg or 1200mg ASP2151 on Days 1 and 7, 100 mg ciclosporin twice daily on Days 3-9, and once in the morning of Day 10. Two participants were withdrawn during the washout period, in the second intervention, another participants were replaced.
Groups:
- ASP2151 400mg: "ASP2151 400mg followed by ASP2151 400mg + 100mg ciclosporin" first, then "ASP and 1200mg mg followed by ASP2151 1200mg + 100mg ciclosporin"
- ASP2151 1200mg: "ASP2151 1200mg followed by ASP2151 1200mg + 100mg ciclosporin" first, then "ASP and 400mg mg followed by ASP2151 400mg + 100mg ciclosporin"
Period: First Intervention(2 Weeks)
Arm/Group | ASP2151 400mg | ASP2151 1200mg
Started | 12 | 12
Received Intervention | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | ASP2151 400mg | ASP2151 1200mg
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention(2 Weeks)
Arm/Group | ASP2151 400mg | ASP2151 1200mg
Started | 12 | 12
Received Intervention | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASP2151 400mg | ASP2151 1200mg | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 33.6 (7.4) | 31.8 (7.1) | 32.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of ASP2151
Time Frame: prior to initial dose on Day 1 and 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36 and 48 h after ASP2151 dosing on Day 1 and Day 7, and also 72 h after ASP2151 dosing on Day 7.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- ASP2151 400mg Alone: ASP2151(400mg) alone
- ASP2151 400mg With Ciclosporin: ASP2151 400mg + 100mg ciclosporin
  ASP2151 400mg + 100mg ciclosporin
- ASP2151 1200mg Alone: ASP2151(1200mg) alone
- ASP2151 1200mg With Ciclosporin: ASP2151 1200mg + 100mg ciclosporin
  ASP2151 1200mg + 100mg ciclosporin
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 1818.0 (26.1) | 1202.3 (31.5) | 3573.1 (26.1) | 2452.1 (31.4)

2. Primary Outcome: Time of Peak Concentration (Tmax) of ASP2151
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 3.00 [0.50 to 4.02] | 4.00 [1.00 to 8.00] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 8.00]

3. Primary Outcome: Area Under the Curve (AUC) of ASP2151
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 23307.4 (27.1) | 19013.5 (31.4) | 48051.2 (25.0) | 37940.8 (25.9)

4. Primary Outcome: Half-Life (t1/2) of ASP2151
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 7.755 (12.1) | 8.593 (16.4) | 7.457 (13.2) | 8.326 (14.1)

5. Primary Outcome: Apparent Total Body Clearance (CL/F) of ASP2151 From Plasma
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
L/h | 17.745 (4.6288) | 21.917 (5.9182) | 25.695 (6.3004) | 32.699 (9.3284)

6. Primary Outcome: Apparent Volume of Distribution (Vd/F) of ASP2151
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
L | 196.9 (45.72) | 269.6 (69.57) | 276.5 (69.55) | 395.3 (118.47)

7. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Refer to the result of adverse event.
Time Frame: Up to 31 days after the Day 7 dose of ASP2151
Measure: Number; unit: participants
Groups:
- 400 mg ASP Treatment: 400 mg ASP Treatment
- 1200 mg ASP Treatment: 1200 mg ASP Treatment
Arm/Group | 400 mg ASP Treatment | 1200 mg ASP Treatment
Number analyzed (Participants) | 24 | 24
participants
  Non-serious adverse event | 15 | 15
  serious adverse event | 0 | 0

8. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of ASP1955888-00
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 173.0 (35.2) | 132.6 (28.1) | 387.3 (38.1) | 307.2 (42.7)

9. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of AS195588-00
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 3.03 [1.00 to 6.00] | 4.00 [3.00 to 8.08] | 3.53 [2.00 to 4.00] | 4.00 [3.00 to 6.02]

10. Other Pre Specified Outcome: Area Under the Curve (AUC) of AS195588-00
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 2614.4 (27.4) | 2441.3 (20.2) | 6147.4 (29.7) | 5584.5 (31.0)

11. Other Pre Specified Outcome: Half-Life (t1/2) of AS195588-00
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | ASP2151 400mg Alone | ASP2151 400mg With Ciclosporin | ASP2151 1200mg Alone | ASP2151 1200mg With Ciclosporin
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 8.59 (15.3) | 9.62 (18.4) | 8.25 (14.3) | 9.02 (16.4)

12. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of Ciclosporin
Time Frame: Blood samples were taken at pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 after dosing of ciclosporin on Days 6 and 7.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Ciclosporin After ASP2151(400mg): Ciclosporin after ASP2151(400mg)
- Ciclosporin With ASP2151(400mg): Ciclosporin with ASP2151(400mg)
- Ciclosporin After ASP2151(1200mg): Ciclosporin after ASP2151(1200mg)
- Ciclosporin With ASP2151(1200mg): Ciclosporin with ASP2151(1200mg)
Arm/Group | Ciclosporin After ASP2151(400mg) | Ciclosporin With ASP2151(400mg) | Ciclosporin After ASP2151(1200mg) | Ciclosporin With ASP2151(1200mg)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 491.0 (18.6) | 482.3 (18.3) | 467.0 (23.7) | 440.0 (18.6)

13. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of Ciclosporin
Time Frame: as for outcome 12
Measure: Median (Full Range); unit: h
Arm/Group | Ciclosporin After ASP2151(400mg) | Ciclosporin With ASP2151(400mg) | Ciclosporin After ASP2151(1200mg) | Ciclosporin With ASP2151(1200mg)
Number analyzed (Participants) | 24 | 24 | 24 | 24
h | 2.00 [1.00 to 3.00] | 2.00 [0.92 to 3.00] | 2.00 [1.00 to 3.00] | 2.00 [0.98 to 4.00]

14. Other Pre Specified Outcome: Area Under the Curve (AUC) of Ciclosporin
Time Frame: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ciclosporin After ASP2151(400mg) | Ciclosporin With ASP2151(400mg) | Ciclosporin After ASP2151(1200mg) | Ciclosporin With ASP2151(1200mg)
Number analyzed (Participants) | 24 | 24 | 24 | 24
h*ng/mL | 1944.3 (19.7) | 2011.0 (22.1) | 1894.2 (22.9) | 1888.2 (19.6)

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- ASP2151(400mg) Alone: Participants who administered ASP2151 alone during the treatment session 1(ASP2151 400mg)
- Ciclosporin After ASP2151(400mg): Participants who administered ciclosporin alone during the treatment session 1(ASP2151 400mg)
- Ciclosporin With ASP2151(400mg): Participants who coadministered ciclosporin and ASP2151during the treatment session 1(ASP2151 400mg)
- ASP2151(1200mg) Alone: Participants who administered ASP2151 alone during the treatment session 1(ASP2151 1200mg)
- Ciclosporin After ASP2151(1200mg): Participants who administered ciclosporin alone during the treatment session 1(ASP2151 1200mg)
- Ciclosporin With ASP2151(1200mg): Participants who coadministered ciclosporin and ASP2151during the treatment session 1(ASP2151 1200mg)
Arm/Group | ASP2151(400mg) Alone | Ciclosporin After ASP2151(400mg) | Ciclosporin With ASP2151(400mg) | ASP2151(1200mg) Alone | Ciclosporin After ASP2151(1200mg) | Ciclosporin With ASP2151(1200mg)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 5/24 | 10/24 | 3/24 | 3/24 | 11/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASP2151(400mg) Alone (N=24) | Ciclosporin After ASP2151(400mg) (N=24) | Ciclosporin With ASP2151(400mg) (N=24) | ASP2151(1200mg) Alone (N=24) | Ciclosporin After ASP2151(1200mg) (N=24) | Ciclosporin With ASP2151(1200mg) (N=24)
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Influenza-like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No